CLINICAL TRIAL: NCT03907358
Title: The Pathogenesis of Age-related Cataract
Brief Title: The Pathogenesis of Human Senile Cataract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Haidong Zou, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Shanghai1st-cataract-001
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cataract in old age
  Interventions: Procedure: phacoemulsification
- cataract in young age
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification

SUMMARY:
To study the pathological mechanism of cataract by genomics, transcriptomics, and proteomics.

DETAILED DESCRIPTION:
Tissue samples and aqueous humor samples will be collected from each individual patients by cataract surgery. After sample treatment, different techniques will be applied for analysis. And bioinformatics approach is applied for data treatment and analysis.The data of genomics, transcriptomics, and proteomics will be analyzed for study of pathological mechanism of cataract.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the explicit diagnosis of cataract (including senile cataract, congenital cataract, complicated cataract, metabolic cataract, traumatic cataract, etc.) in the operated eye are willing to undergo cataract surgery.

Exclusion Criteria:

* Patients whose cataracts need not be operated
* Patients with any contraindications to cataract surgery
* Patients are unwilling to undergo cataract surgery

Ages: 5 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the explicit diagnosis of cataract are willing to undergo cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-12-07 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Characterization of miRNA in micro-scale human aqueous humor | 12 month
  method development for miRNA detection in aqueous humor
Favored amplification recovery via protection-chromatin immunoprecipitation-Seq of human eye tissue samples | 24 month
  low-cell-number epigenome profiling for study of cataract
Study of cataract by genomics, transcriptomics, and proteomics approaches | 36 month
  detect histone H3 lysine 4 trimethylation (H3K4me3) of aqueous humor of cataract patients by genomics, transcriptomics, and proteomics methods

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Shanghai General Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided